CLINICAL TRIAL: NCT01334034
Title: A Trial Investigating the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of NNC 0123-0000-0338 in Healthy Subjects
Brief Title: Safety of NNC 0123-0000-0338 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN1953-3832; U1111-1118-2525 (Other: WHO); 2010-023885-38 (EudraCT Number)
Record Dates: First submitted 2011-04-11; First posted 2011-04-12 (Estimated); Last update posted 2017-03-01 (Actual); Status verified 2017-02

CONDITIONS: Diabetes; Healthy
MeSH Terms: conditions — Diabetes Mellitus | interventions — Insulin Glargine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dose levels 1-7 (Experimental)
  Interventions: Drug: NNC 0123-0000-0338; Drug: placebo; Drug: insulin glargine

INTERVENTIONS:
Drug: NNC 0123-0000-0338 — Subjects will be randomised to receive a single dose of NNC 0123-0000-0338 (tablet), at 7 escalating dose levels. Progression to next dose level will be based on a safety evaluation.
Drug: placebo — Subjects will receive a single dose of placebo (tablet), as a comparator to NNC 0123-0000-0338 at all dose levels. Placebo dose remains the same at all dose levels.
Drug: insulin glargine — As an open label active comparator, a single dose of insulin glargine will be administered subcutaneously (under the skin), at all dose levels. Insulin glargine dose remains the same at all dose levels.

SUMMARY:
This trial is conducted in Europe. The aim of this trial is to investigate the safety, tolerability, pharmacokinetics (the exposure of the trial drug in the body), and the pharmacodynamics (the effect of the investigated drug on the body) of NNC 0123-0000-0338 as tablets in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Male subject
* Body mass index (BMI) between 18 and 28 kg/m^2 (both inclusive)

Exclusion Criteria:

* Known or suspected hypersensitivity to trial products or related products
* Presence of clinically significant acute gastrointestinal symptoms (e.g. nausea, vomiting, heartburn or diarrhoea) within 2 weeks prior to dosing, as judged by the trial physician
* Presence of any medical condition that may confound the results of the trial or pose an unacceptable risk to the subject by administering the trial product, as judged by the trial physician

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2011-04-11 (Actual); Primary Completion 2011-09-16 (Actual); Study Completion 2011-09-16 (Actual)

PRIMARY OUTCOMES:
Number of adverse events | from trial product administration and until completion of the dosing visit (Day 0 to Day 6)

SECONDARY OUTCOMES:
Area under the serum insulin concentration-time curve | from 0 to 120 hours after a single dose
Area under the glucose infusion rate-time curve | from 0 to 24 hours after a single dose

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Neuss, Germany

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com